CLINICAL TRIAL: NCT00596479
Title: Subcutaneous Delivery of Filgrastim (rG-CSF) for the Promotion of Collateral Growth in Patients With Coronary Artery Disease
Brief Title: Filgrastim for the Promotion of Collateral Growth in Patients With CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05/04
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease
Keywords: CAD; G-CSF; Collaterals; CFI; perfusion
MeSH Terms: conditions — Coronary Artery Disease | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Filgrastim (rG-CSF)

SUMMARY:
The purpose of this study in humans with stable coronary artery disease (CAD) treatable by PCI (percutaneous coronary intervention) is to evaluate the safety and efficacy of subcutaneous delivery of recombinant granulocyte colony stimulating factor rG-CSF (Filgrastim, Neupogen®, Amgen Switzerland) with regard to the promotion of collateral growth.

DETAILED DESCRIPTION:
The purpose of this study in humans with stable coronary artery disease (CAD) treatable by PCI (percutaneous coronary intervention) is to evaluate the safety and efficacy of subcutaneous delivery of recombinant granulocyte colony stimulating factor rG-CSF (Filgrastim, Neupogen®, Amgen Switzerland) with regard to the promotion of collateral growth.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* 1- to 3-vessel coronary artery disease (CAD)
* Stable angina pectoris
* At least 1 stenotic lesion suitable for PCI
* No Q-wave myocardial infarction in the area undergoing CFI measurement
* Written informed consent to participate in the study

Exclusion Criteria:

* Patients admitted as emergencies
* Acute myocardial infarction
* Unstable CAD
* CAD treated best by CABG
* Patients with overt neoplastic disease
* Patients with diabetic retinopathy
* Liver or kidney disease
* Pre-menopausal women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Collateral flow index (CFI) at 2 weeks follow-up compared to baseline CFI

SECONDARY OUTCOMES:
Absolute myocardial perfusion during hyperemia by contrast echocardiography (MCE) at baseline, at 2 weeks and at 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Gloekler, MD, Principal Investigator — University of Bern; Tobias Rutz, MD, Principal Investigator — University of Bern; Pascal Meier, MD, Principal Investigator — University of Bern; Christian Seiler, MD, Study Chair — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Meier P, Gloekler S, de Marchi SF, Indermuehle A, Rutz T, Traupe T, Steck H, Vogel R, Seiler C. Myocardial salvage through coronary collateral growth by granulocyte colony-stimulating factor in chronic coronary artery disease: a controlled randomized trial. Circulation. 2009 Oct 6;120(14):1355-63. doi: 10.1161/CIRCULATIONAHA.109.866269. Epub 2009 Sep 21. PMID 19770393